CLINICAL TRIAL: NCT06289413
Title: Autonomic Dysfunction in Patients Following Bariatric Surgery: The ADiPOSE Study
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart and Rhythm Institute, Overland Park, KS (Unknown); Bariatric and Metabolic Specialists, Overland Park, KS (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_ADiPOSE_0027
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Autonomic Dysfunction; Orthostatic Intolerance
MeSH Terms: conditions — Primary Dysautonomias; Orthostatic Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Development of AD/OI after BS.
  Interventions: Other: Development of AD/OI after BS

INTERVENTIONS:
Other: Development of AD/OI after BS — OI is a type of AD that results in chronic supine-to-standing hypotension and disabling dizziness, lightheadedness, and even syncope. Whether arising from malabsorption, vagus nerve damage, or splanchnic vasodilation, the pathophysiology of OI in bariatric surgery is not clear and requires more investigation.
  Treatment of OI usually consists of dietary and lifestyle changes, which may include compression stockings and abdominal binders. Medical options include peripheral vasoconstrictors and mineralocorticoids; some patients may be referred to Cardiology for further testing. Management is difficult and endurance and tilt training, inflatable abdominal bands, and beta-blockers have been proposed. One recent study demonstrated the treatment of refractory OI with Droxidopa. Yet, the success of treatment is individualized and necessitates more novel approaches.

SUMMARY:
Observational two phase, retrospective and prospective registry study to assess the prevalence of and characterize outcomes of autonomic dysfunction (AD) in patients who undergo bariatric surgery (BS) and to better define the underlying pathophysiology of AD following BS.

DETAILED DESCRIPTION:
Previous studies have investigated the incidence of OI (orthostatic intolerance) with BS. One recent meta-analysis only found a 5-year cumulative incidence of 4.2%, challenging reports of increased incidence. However, this same study recognized the limited and low-quality evidence investigating this phenomenon. Other meta-analyses found only four studies each that matched their search criteria, highlighting the lack of evidence. Thus, this study is designed to investigate the prevalence and better understand AD/OI after BS.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 - 85 years
* Can provide consent
* Negative urine B-hCG
* Continued follow-up with the bariatric surgery team.
* BS includes one of the following: gastric bypass, sleeve gastrectomy, and biliopancreatic diversion with duodenal switch.
* Phase I: Underwent BS within the last 3 years
* Phase II: Will undergo BS within the next 3 months or underwent BS in the last 30 days

Exclusion Criteria:

* Unable to provide consent
* Pregnant or breastfeeding
* BMI < 35
* Revision surgery of one of the following BS from above
* Prior history of autonomic dysfunction prior to BS
* Developed AD 72 months post-procedure
* No evidence of AD/OI

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Phase I: who have undergone bariatric surgery in the last 3 years. Phase II: who will undergo bariatric surgery within the next 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of and characterize outcome of autonomic dysfunction (AD) in patients who undergo bariatric surgery (BS) | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (8):
- United States (8):
  - Menorah Medical Center, Overland Park, Kansas
  - Bariatric and Metabolic Specialists, Overland Park, Kansas
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lazzati A. Epidemiology of the surgical management of obesity. J Visc Surg. 2023 Apr;160(2S):S3-S6. doi: 10.1016/j.jviscsurg.2022.12.004. Epub 2023 Jan 30. PMID 36725453
- [Background] Arterburn DE, Telem DA, Kushner RF, Courcoulas AP. Benefits and Risks of Bariatric Surgery in Adults: A Review. JAMA. 2020 Sep 1;324(9):879-887. doi: 10.1001/jama.2020.12567. PMID 32870301
- [Background] Zhang JB, Tamboli RA, Albaugh VL, Williams DB, Kilkelly DM, Grijalva CG, Shibao CA. The incidence of orthostatic intolerance after bariatric surgery. Obes Sci Pract. 2019 Dec 6;6(1):76-83. doi: 10.1002/osp4.383. eCollection 2020 Feb. PMID 32128245
- [Background] Rodriguez Ruben, J., et al., AUTONOMIC DYSFUNCTION FOLLOWING BARIATRIC SURGERY. Journal of the American College of Cardiology, 2021. 77(18_Supplement_1): p. 327-327
- [Background] Tanaka H, Yamaguchi H, Tamai H. Treatment of orthostatic intolerance with inflatable abdominal band. Lancet. 1997 Jan 18;349(9046):175. doi: 10.1016/S0140-6736(97)24003-1. No abstract available. PMID 9111544
- [Background] Ector H, Reybrouck T, Heidbuchel H, Gewillig M, Van de Werf F. Tilt training: a new treatment for recurrent neurocardiogenic syncope and severe orthostatic intolerance. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 2):193-6. doi: 10.1111/j.1540-8159.1998.tb01087.x. PMID 9474671
- [Background] Freitas J, Santos R, Azevedo E, Costa O, Carvalho M, de Freitas AF. Clinical improvement in patients with orthostatic intolerance after treatment with bisoprolol and fludrocortisone. Clin Auton Res. 2000 Oct;10(5):293-9. doi: 10.1007/BF02281112. PMID 11198485
- [Background] Winker R, Barth A, Bidmon D, Ponocny I, Weber M, Mayr O, Robertson D, Diedrich A, Maier R, Pilger A, Haber P, Rudiger HW. Endurance exercise training in orthostatic intolerance: a randomized, controlled trial. Hypertension. 2005 Mar;45(3):391-8. doi: 10.1161/01.HYP.0000156540.25707.af. Epub 2005 Feb 7. PMID 15699447
- [Background] Kokorelis C, Bodurtha J, Guthrie K, Rowe PC. Successful Treatment of Refractory Orthostatic Intolerance (OI) With Droxidopa. Clin Pediatr (Phila). 2022 Oct;61(9):593-595. doi: 10.1177/00099228221092645. Epub 2022 Jun 8. No abstract available. PMID 35678018
- [Background] Al Nou'mani J, Al Alawi AM, Falhammar H, Al Qassabi A. Orthostatic intolerance after bariatric surgery: A systematic review and meta-analysis. Clin Obes. 2021 Dec;11(6):e12483. doi: 10.1111/cob.12483. Epub 2021 Aug 19. PMID 34409762
- [Background] Kermansaravi M, Chiappetta S, Lainas P, Kassir R. Orthostatic Intolerance after Bariatric Surgery: a Systematic Review. Obes Surg. 2021 May;31(5):2250-2254. doi: 10.1007/s11695-021-05266-4. Epub 2021 Mar 2. PMID 33655427
- [Background] Addison P, Carsky K, Patti ME, Roslin M. Hypoglycemia and Dysautonomia After Bariatric Surgery: a Systematic Review and Perspective. Obes Surg. 2022 May;32(5):1681-1688. doi: 10.1007/s11695-022-05960-x. Epub 2022 Feb 8. PMID 35133603
- [Background] Honka H, Koffert J, Kauhanen S, Teuho J, Hurme S, Mari A, Lindqvist A, Wierup N, Groop L, Nuutila P. Bariatric Surgery Enhances Splanchnic Vascular Responses in Patients With Type 2 Diabetes. Diabetes. 2017 Apr;66(4):880-885. doi: 10.2337/db16-0762. Epub 2017 Jan 17. PMID 28096259
- [Background] Hatipoglu S, Akbulut S, Hatipoglu F, Abdullayev R. Effect of laparoscopic abdominal surgery on splanchnic circulation: historical developments. World J Gastroenterol. 2014 Dec 28;20(48):18165-76. doi: 10.3748/wjg.v20.i48.18165. PMID 25561784
- [Background] Williams WH 3rd, Browne RC, Bui TP, Holmes AA, Thakar D. Case report on intravenous octreotide for the treatment of intraoperative vasoplegia following thymoma resection. SAGE Open Med Case Rep. 2019 Feb 8;7:2050313X19827744. doi: 10.1177/2050313X19827744. eCollection 2019. PMID 30800305
- [Background] Chan MM, Chan MM, Mengshol JA, Fish DN, Chan ED. Octreotide: a drug often used in the critical care setting but not well understood. Chest. 2013 Dec;144(6):1937-1945. doi: 10.1378/chest.13-0382. PMID 24297127
- [Background] Chatila R, Ferayorni L, Gupta T, Groszmann RJ. Local arterial vasoconstriction induced by octreotide in patients with cirrhosis. Hepatology. 2000 Mar;31(3):572-6. doi: 10.1002/hep.510310304. PMID 10706544
- [Background] Karwa R, Woodis CB. Midodrine and octreotide in treatment of cirrhosis-related hemodynamic complications. Ann Pharmacother. 2009 Apr;43(4):692-9. doi: 10.1345/aph.1L373. Epub 2009 Mar 18. PMID 19299324